CLINICAL TRIAL: NCT07352293
Title: The Value of Using Methotrexate Therapy Along With Non Cultured Epidermal Cell Suspension (NCES) in Stable Resistant Vitiligo: An Interventional Prospective Randomized Controlled Trial.
Brief Title: The Value of Methotrexate in NCES for Stable Vitiligo
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nanis Aleem Abdul Moneim Ragab, Associate professor of Dermatology Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTXNCES
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Vitiligo
Keywords: Methotrexate; NCES; acral vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCES (Active Comparator)
  Interventions: Procedure: Non cultured epidermal suspension
- NCES+Methotexate (Experimental)
  Interventions: Procedure: Non cultured epidermal suspension

INTERVENTIONS:
Procedure: Non cultured epidermal suspension — Under aseptic precautions and local anesthesia, a Thiersch graft about one-third the size of the recipient area will be harvested from the donor site (usually upper thigh/ buttocks). The skin graft will be transferred to trypsin-EDTA solution and incubated at 37 °C for 20-30 minutes to separate epidermis from the dermis and then washed with PBS. The tissue will be teased gently with sterile forceps to release epidermal cells from the trypsin digested graft. The white dermis will be removed, and the suspension will be centrifuged at 1000g for 5-10 minutes and the supernatant will be discarded.
  Under strict asepsis, the recipient vitiliginous areas will be anesthetized followed by fractional laser CO2 resurfacing, using dot mode off resurfacing at a power of 18-20 W, dwell time 1,500-2000 milliseconds (DEKA, Florence, Italy). One to three passes will be performed until the epidermis is removed uniformly. Then, the NCES will be applied and uniformly spread.

SUMMARY:
The goal of this clinical trial is to learn if adding a six months course of Methotrexate would improve the results of non cultured epidermal suspension (NCES) in adult patients with acral and resistant vitiligo lesions over the elbows and knees. researchers will compare results of NCES in two groups one group will receive Methotrexate for 3 months prior to the procedure and 3 months after the procedure, while the other group will not receive the drug. Patients will receive PUVA hand & feet 3 times/week for 3 months after NCES during this period they will be followed up monthly to evaluate repigmentation.

DETAILED DESCRIPTION:
Depending on the type, extent, and duration of vitiligo, conventional medical therapies such as topical and systemic corticosteroids, topical immunomodulators, and phototherapy are not always successful, and repigmentation is often incomplete. Acral vitiligo as well as vitiligo over friction sites as elbows and knees are resistant to treatment including surgical procedures. Relatively less melanocyte density as well as higher chances of koebnerization over these friction and injury prone anatomical sites were among the suggestions for poor response to treatment. It was also found that melanocyte growth and migration in acral vitiligo is hindered by several factors such as decreased MMP9, MMP2, c-kit and MHCII expression, together with higher expression of antimelanogenic factors as tenascin and DKK1. Non-cultured epidermal cellular suspension (NCES) is a cellular grafting technique, whose major advantage is permitting treatment of affected skin surface area up to 10 times larger than the donor area without culturing. Methotrexate is an antifolate drug, that decreases the number of T cells. Studies showed that methotrexate has a positive effect on the stabilization of vitiligo. Combined treatment with phototherapy allows better and faster repigmentation than phototherapy alone. Systemic drugs have been previously used perioperatively in vitiligo surgery. Oral betamethasone has been previously used in the peri surgical period and was reported to increase the chances of complete repigmentation in large vitiliginous lesions as activity at the cellular level is still plausible in spite of clinical stability. The aim of this study is to assess whether adding methotrexate therapy to NCES in the peri surgical period would improve repigmentation in acral vitiligo and other resistant sites.

* Inclusion criteria:

  * Patients with non-segmental vitiligo (NSV) with acral or resistant lesions over the elbows and knees, that has not responded to conventional treatment
  * Stability for ≥ 1 year
  * Age ≥18 years
  * Lack of topical treatment for at least 1 month prior to surgery and systemic treatment for at least 3 months prior to surgery.
* Exclusion criteria:

  * Non acral NSV responsive to conventional treatment modalities
  * Active vitiligo; new lesions, expansion of old lesions, confetti like lesions, ill-defined edges or koebnerization in < 1 year
  * Age < 18 years.
  * Pregnant females.
  * Patients with hematologic, hepatic, renal disease or chronic infection.
  * Topical treatment in the past month and systemic treatment in the past 3 months.
* Methodology in details:
* forty lesions in patients with stable vitiligo will be recruited (20 size and region matched lesions per group). An informed written consent will be obtained from patients.
* Patients will be randomized using a computer generated list to one of the two groups which are age and sex matched:

Group A will undergo None cultured epidermal suspension (NCES) without methotrexate.

Group B will receive methotrexate 15 mg/week for 3 months prior to NCES and for 3 months afterwards.

Clinical assessment:

Baseline assessment will include assessing any pigmentation within the patch to be transplanted using the VESTA score and its surface area using point counting technique.

Standardized photographs will be taken at initial assessment, and by the end of the study period after 3 months.

Under aseptic precautions and local anesthesia, a Thiersch graft about one-third the size of the recipient area will be harvested from the donor site (usually upper thigh/ buttocks). The skin graft will be transferred to trypsin-EDTA solution and incubated at 37 °C for 20-30 minutes to separate epidermis from the dermis and then washed with PBS. The tissue will be teased gently with sterile forceps to release epidermal cells from the trypsin digested graft. The white dermis will be removed, and the suspension will be centrifuged at 1000g for 5-10 minutes and the supernatant will be discarded.

Under strict asepsis, the recipient vitiliginous areas will be anesthetized followed by fractional laser CO2 resurfacing, using dot mode off resurfacing at a power of 18-20 W, dwell time 1,500-2000 milliseconds (DEKA, Florence, Italy). One to three passes will be performed until the epidermis is removed uniformly. Then, the NCES will be applied and uniformly spread. It will be covered with a dry collagen sheet followed by sterile surgical pad and tegaderm.

The area will be immobilized after bandaging and the patient will be advised to restrict movement at the operated site.

Patients will start a 1-week course of antibiotics. Dressings will be removed after 1 week, and patients will start topical PUVA hand and feet, 3 times per week for 3 months.

Patients will be followed up monthly for 3 months following the first visit at 1 week.

Both qualitative and quantitative assessment will be done after 3 months of PUVA Hand and feet. Qualitatively, blinded physician assessment of repigmentation as well as color match will be done based on baseline photographs. Quantitatively, point counting method as well as VESTA score will be used as well to assess the surface area of the residual depigmented area and degree of repigmentation respectively.

ELIGIBILITY:
* Inclusion criteria:

  * Patients with non-segmental vitiligo (NSV) with acral or resistant lesions over the elbows and knees, that has not responded to conventional treatment
  * Stability for ≥ 1 year
  * Age ≥18 years
* Exclusion criteria:

  * Segmental vitiligo
  * Active vitiligo; new lesions, expansion of old lesions, confetti like lesions, ill-defined edges or koebnerization in < 1 year
  * Age < 18 years.
  * Pregnant females.
  * Patients with hematologic, hepatic, renal disease or chronic infection.
  * Topical treatment in the past month and systemic treatment in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent change in surface area by point counting method after NCES alone versus NCES combined with MTX | 3 months
  A decrease in the surface area (number of points) of depigmented area indicates successful regimentation
Percent change in surface area by VESTA score after NCES alone versus NCES combined with MTX | 3 months
  VESTA score ranges between 0-100% (0 % is complete depigmentation and 100% is fully pigmented) an increase in VESTA score indicates successful regimentation

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Outpatient Clinic, Kasr al Ainy Teaching Hospital, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
I will share the deidentified data sheet of the results of the trial
Supporting Information: Study Protocol, SAP
Time Frame: 1 month after paper publication

REFERENCES:
- [Background] Tavitova A, Valle Y, Lomonosov K. Using methotrexate in the treatment of advanced vitiligo. J Cosmet Dermatol. 2023 Mar;22(3):1136-1138. doi: 10.1111/jocd.15524. Epub 2022 Nov 21. No abstract available. PMID 36409563
- [Background] Alghamdi K, Khurrum H. Methotrexate for the treatment of generalized vitiligo. Saudi Pharm J. 2013 Oct;21(4):423-4. doi: 10.1016/j.jsps.2012.12.003. No abstract available. PMID 24227963
- [Background] Seneschal J, Speeckaert R, Taieb A, Wolkerstorfer A, Passeron T, Pandya AG, Lim HW, Ezzedine K, Zhou Y, Xiang F, Thng S, Tanemura A, Suzuki T, Rosmarin D, Rodrigues M, Raboobee N, Pliszewski G, Parsad D, Oiso N, Monteiro P, Meurant JM, Maquignon N, Lui H, Le Poole C, Leone G, Lee AY, Lan E, Katayama I, Huggins R, Oh SH, Harris JE, Hamzavi IH, Gupta S, Grimes P, Goh BK, Ghia D, Esmat S, Eleftheriadou V, Bohm M, Benzekri L, Bekkenk M, Bae JM, Alomar A, Abdallah M, Picardo M, van Geel N. Worldwide expert recommendations for the diagnosis and management of vitiligo: Position statement from the international Vitiligo Task Force-Part 2: Specific treatment recommendations. J Eur Acad Dermatol Venereol. 2023 Nov;37(11):2185-2195. doi: 10.1111/jdv.19450. Epub 2023 Sep 15. PMID 37715487
- [Background] Karagaiah P, Valle Y, Sigova J, Zerbinati N, Vojvodic P, Parsad D, Schwartz RA, Grabbe S, Goldust M, Lotti T. Emerging drugs for the treatment of vitiligo. Expert Opin Emerg Drugs. 2020 Mar;25(1):7-24. doi: 10.1080/14728214.2020.1712358. Epub 2020 Feb 3. PMID 31958256
- [Background] Silpa-Archa N, Griffith JL, Huggins RH, Henderson MD, Kerr HA, Jacobsen G, Mulekar SV, Lim HW, Hamzavi IH. Long-term follow-up of patients undergoing autologous noncultured melanocyte-keratinocyte transplantation for vitiligo and other leukodermas. J Am Acad Dermatol. 2017 Aug;77(2):318-327. doi: 10.1016/j.jaad.2017.01.056. Epub 2017 May 11. PMID 28502377
- [Background] Esmat S, Assaf MI, Mohye Eldeen R, Gawdat HI, Saadi DG. Evaluation of needling/microneedling as an adjunct to phototherapy in the treatment of stable acral vitiligo: a comparative clinical and immunohistochemical study. J Dermatolog Treat. 2022 Aug;33(5):2621-2628. doi: 10.1080/09546634.2022.2062279. Epub 2022 Apr 8. PMID 35373693
- [Background] Abdel Halim DM, Fekry A, Mogawer RM. The value of adding platelet-rich plasma (PRP) to noncultured epidermal cell suspension (NCECS) in surgical treatment of stable resistant vitiligo: A self-controlled randomised double-blinded study. Australas J Dermatol. 2023 Aug;64(3):359-367. doi: 10.1111/ajd.14080. Epub 2023 May 25. PMID 37228170
- [Background] Huggins RH, Henderson MD, Mulekar SV, Ozog DM, Kerr HA, Jabobsen G, Lim HW, Hamzavi IH. Melanocyte-keratinocyte transplantation procedure in the treatment of vitiligo: the experience of an academic medical center in the United States. J Am Acad Dermatol. 2012 May;66(5):785-93. doi: 10.1016/j.jaad.2011.05.002. Epub 2011 Aug 23. PMID 21864935
- [Background] Esmat SM, El-Tawdy AM, Hafez GA, Zeid OA, Abdel Halim DM, Saleh MA, Leheta TM, Elmofty M. Acral lesions of vitiligo: why are they resistant to photochemotherapy? J Eur Acad Dermatol Venereol. 2012 Sep;26(9):1097-104. doi: 10.1111/j.1468-3083.2011.04215.x. Epub 2011 Aug 18. PMID 21851425
- [Background] Falabella R. Surgical approaches for stable vitiligo. Dermatol Surg. 2005 Oct;31(10):1277-84. doi: 10.1111/j.1524-4725.2005.31203. PMID 16188179
- [Background] Mulekar SV. Stable vitiligo treated by a combination of low-dose oral pulse betamethasone and autologous, noncultured melanocyte-keratinocyte cell transplantation. Dermatol Surg. 2006 Apr;32(4):536-41. doi: 10.1111/j.1524-4725.2006.32109.x. PMID 16681662